CLINICAL TRIAL: NCT01959581
Title: An Innovative Device for Intervention in Infants With Nervous System Injury
Brief Title: Movement Enhancing Device for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Christiana Care Health Services (Other); Alfred I. duPont Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD076092-01A1 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Upper Extremity Dysfunction
Keywords: Wilmington Robotic Exoskeleton; Reaching; Upper extremity function; Preterm Infants; Brain injury; Pediatrics; Early Intervention; Arthrogryposis
MeSH Terms: conditions — Brain Injuries; Arthrogryposis

STUDY DESIGN:
Masking Description: Coders are blind to which study phase participants are in
Oversight: Data Monitoring Committee: No

ARMS (1):
- Movement enhancing device (Other): Guided play while wearing a movement assisting device
  Interventions: Device: Movement Enhancing Device

INTERVENTIONS:
Device: Movement Enhancing Device — Naturalistic play activities using the hands while wearing the movement enhancing device.
  Other Names: WREX (Wilmington Robotic Exoskeleton)

SUMMARY:
The purpose of this study is to assess: 1) how infants move their bodies to explore, play, and solve problems, 2) if this is different in a high-risk group of infants, and 3) if these abilities can be advanced in a high-risk group through the use of a movement assisting device.

DETAILED DESCRIPTION:
Certain conditions or diagnoses identified soon after birth are known to put infants at risk for having problems with their motor (movement) development as they get older. Infants with these diagnoses are at risk for additional developmental problems due to their inability to move their bodies to explore, learn, and play. This study tests how a device that assists movement can help exploration, learning, and play in children. The information gathered in this study will help us better understand how early learning happens and how we can help individuals become better movers, learners, and problem-solvers so they can increase their participation in everyday play activities.

ELIGIBILITY:
Inclusion Criteria:

• Infants will be invited to participate if they are between 1 month and 6 years and:

* Were born < 36 weeks of gestational age with periventricular leukomalacia or grade III or IV intraventricular hemorrhage
* Were born > 36 weeks of gestational age with encephalopathy related to perinatal asphyxia
* Have the diagnosis of neonatal stroke or intracranial hemorrhage
* Have brachial plexus palsy
* Have arthrogryposis multiplex congenital
* Have Down syndrome
* Have congenital hypotonia

Exclusion Criteria:

• blindness or severe sensory motor impairments that would prohibit the child from completing the study assessment.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele A Lobo, PT, PhD, Principal Investigator — University of Delaware
Locations (3):
- United States (3):
  - Christiana Care Health Services, Newark, Delaware
  - University of Delaware, Newark, Delaware
  - Nemours Foundation, Wilmington, Delaware

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Movement Enhancing Device
Started | 30
Completed | 25
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Movement Enhancing Device
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.37 (1.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Time Contacting Objects
Description: Percent of the assessment time participants are able to contact objects across different locations. Change within each session with versus without the exoskeleton donned. Slope of change across time in the intervention phase relative to in the baseline phase.
Time Frame: 7 months
Population: infants born with significant brain injury and toddlers with a diagnosis of arthrogryposis multiplex congenita
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Movement Enhancing Device
Number analyzed (Participants) | 20
percentage of time | 40.75 (30.06)
Statistical Analysis 1: Comparison: Movement Enhancing Device; Repeated measures ANOVA; Test type: Superiority or Other; p < .05, ANOVA

ADVERSE EVENTS:
Arm/Group | Movement Enhancing Device
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No